CLINICAL TRIAL: NCT07348809
Title: The Effects Of Virtual Reality and Stress Ball Application on Pain, Anxiety Levels and Injection Satisfaction in During Insulin Injection in Geriatric Patients With Type 2 Diabetes
Acronym: TYPE 2 DİABETE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, ezgi mutluay yayla, Principal investigator, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBF.23.004
Record Dates: First submitted 2025-11-26; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diabete Type 2; Virtual Reality; Stress Ball; Procedural Anxiety; Pain Management
Keywords: anxiety; needle; pain; stress ball; Type 2 diabetes; virtual reality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Agnosia; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial with control and intervention groups, pre-test and post-test.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): First, the State-Trait Anxiety Inventory (STAI) was administered as a pre-test before both blood sugar measurement and insulin injection. These procedures were then performed. After their completion, the VAS and STAI were administered again as a post-test
- virtual reality (Experimental): First, the State-Trait Anxiety Inventory (STAI) was administered as a pre-test before blood sugar measurement. Then, five minutes before their blood sugar was taken, patients started watching motivational videos via virtual reality glasses and continued watching throughout the measurement. Before the videos began, patients were given instructions on how to use the headset and what to expect. After the blood sugar measurement, the STAI, VAS and VPSS were administered. Next, the STAI was given as a pre-test before the insulin injection. Five minutes before the insulin injection, motivational videos were again shown through the virtual reality glasses and continued during the injection. Following this procedure, the STAI, VAS, and VPSS were administered once more as a final test.
  Interventions: Device: virtual reality
- stress ball (Experimental): On the second day, the stress ball group's procedures were as follows:
  First, we administered the State-Trait Anxiety Inventory (STAI) as a pre-test before measuring blood sugar levels. Patients were then instructed to focus on and continuously squeeze and release the stress ball until their blood sugar measurement was complete. Afterward, blood sugar measurements were taken. Following the blood sugar measurement, the VAS, STAI and VPSS were administered. Next, the STAI was given as a pre-test before the insulin injection. Patients continued to squeeze and release the stress ball, focusing their attention on it, until the insulin injection was finished. After the injection, the VAS, STAI, and VPSS were administered again as a post-test.
  Interventions: Device: stress ball

INTERVENTIONS:
Device: virtual reality — The patients in the virtual reality group watched motivational videos of their choice from YouTube (e.g., nature scenes, seaside walks, underwater views), accompanied by background music. These videos were displayed using Glasses (featuring a 5.7-inch, 1440x2560 pixel screen resolution display from China) and shown in VR mode via a Samsung A51 smartphone before both blood sugar testing and insulin injection (Figure 1). While previous studies typically showed virtual reality videos for 5-10 minutes (kaynak), in this study, patients viewed motivational videos for 5 minutes to help them more easily immerse themselves in the virtual world.
  Arms: virtual reality
Device: stress ball — The stress balls used in the study were 3 cm in diameter, round, and constructed from medium-hardness, high-quality silicone. These were sourced and distributed to patients by the researchers
  Arms: stress ball

SUMMARY:
The effects of virtual reality and stress ball applied during insulin injection on pain, anxiety levels and injection satisfaction in geriatric patients with type 2 diabetes.

Insulin injection in geriatric patients with type 2 diabetes causes pain and anxiety, making the treatment process difficult. The aim of the study is to determine the effect of virtual reality and stress ball application on pain, anxiety levels and injection satisfaction during insulin injection in geriatric patients with Type 2 diabetes. Randomization will be achieved by randomly and equally distributing patients who meet the sample selection criteria at Tarsus State Hospital to 3 groups (1st experimental group, 2nd experimental group and 3rd group control group) through a computer program. Considering that there may be case losses, a total of 90 patients (1st Experimental Group [virtual reality applied]: 30 patients, 2nd Experimental Group [stress ball applied]: 30 patients, control group: 30 patients) will be included in the sample group. In collecting data; A data collection form consisting of "Personal Information Form", "Visual Analog Scale (VAS)", State Anxiety Inventory (DCI), "Visual Patient Satisfaction Scale" forms will be used.

DETAILED DESCRIPTION:
Diabetes is a disease that occurs due to insufficient production of insulin hormone, deficiency or inability to use the insulin hormone produced. Diabetes is an important disease whose incidence is increasing every year, negatively affecting quality of life and causing morbidity and mortality. According to the 2021 data of the National Diabetes Federation, approximately 10.5% of the adult population worldwide has diabetes and almost half of these patients are not aware of their disease. Type 2 diabetes is the most common form of diabetes and accounts for approximately 90% of the entire population. Many factors such as unfavorable living conditions, low socioeconomic level, obesity and advanced age cause type 2 diabetes. Type 2 diabetes, which is the most common chronic disease seen in geriatric patients and also a serious life-threatening disease, is becoming increasingly common in the elderly population with the prolongation of life expectancy. Aging is a process that leads to many anatomical and physiological changes in individuals and brings with it the risks of various pathological conditions. With this process, there is an increase in the incidence of chronic diseases such as type 2 diabetes, which causes psychological and physiologic decline requiring long-term treatments, close follow-up and serious care. In addition to factors such as lifestyle changes and diabetes awareness, insulin therapy also plays a very important role in the management of diabetes. Insulin treatment is the primary option in case of oral hypoglycemic drug failure or development of diabetes-induced vascular complications. In order to eliminate side effects and have glycemic control in insulin treatment, patients should be knowledgeable about their diseases and insulin treatments, and in addition, they should be competent and have a positive perspective about insulin injection administration. The anxiety experienced by patients during insulin injection may negatively affect emotional well-being and glycemic control. According to the results of a study, it was reported that approximately 48.4% of patients with diabetes experienced noncompliance with treatment because of the pain they would experience during insulin injection and the thought of not being able to endure this pain. In the light of today's technological developments, various methods are applied to patients to divert attention during treatment. Virtual reality and stress ball applications are some of these applications. Thanks to the distraction technique, attention is diverted away from the pain and the severity in the perception of pain is reduced. Nurses play an important role in the management, implementation and rehabilitation of the treatment process of patients. Due to many procedures such as various injection applications, invasive interventions and care applications, nurses are in close interaction with patients and take important responsibilities in the management of many conditions such as pain, fear and anxiety that occur in the patient during this interaction. In some studies in the literature, it is known that virtual reality goggles and stress ball applications are used during dressing changes in patients with burns, painful invasive interventions, chemotherapy applications, bronchoscopy, cystoscopy and hemodialysis. However, there is no study in the literature examining the effect of virtual reality and stress ball applications on pain, anxiety level and injection satisfaction during insulin injection in geriatric patients with type 2 diabetes. This study is thought to contribute to the literature by filling this gap.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or older,
* at least two daily insulin injections and blood sugar monitoring,
* a minimum of 6 months of insulin treatment
* no hand or arm problems preventing stress ball use,
* be able to communicate in Turkish,
* have no orders that would hinder communication (e.g., psychological or related to hearing/understanding)
* volunteer to participate in the study.

Exclusion Criteria:

* if they have: epilepsy, vertigo, anxiety, active nausea, vomiting, or headaches
* regularly use painkillers
* have chronic pain disorders
* have previously experienced virtual reality
* have any problems in the arm's injection area

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Descriptive Information Form were used to collect the data. | The first day;15 minutes before blood sugar measurements and insulin injections are administered
  Descriptive Information Form The descriptive information form was created by evaluating the studies conducted with older adults with type 2 diabetes. A total of 13 questions were asked about the patient's year of birth, education level, marital status, employment status, year of diabetes diagnosis, duration of insulin use, etc. in the descriptive information form.The first day involved no interventional procedures for any group (virtual reality, stress ball, or control). The data collection sequence was as follows: Participants first completed the Descriptive Information Form.
The Visual Patient Satisfaction Scale (VPSS) | The second day; intervention groups were administered after the blood sugar and insulin procedures and after an average of 3-5 minutes.
  This scale, which combines features of the well-known Visual Analogue Scale (VAS), is a 100 mm horizontal line without numbers. It is anchored at one end by 'Not at all satisfied' and at the other by 'Very satisfied.' Patients will use this scale to indicate their level of satisfaction with the virtual reality and stress ball applications by marking the point on the line that best corresponds to their experience. The scale was evaluated and recorded by a nurse who was independent of the study."
Visual analogue scale were used to collect the data. | The first day ; during the blood sugar and insulin procedures and baseline, after an average of 1-2 minutes
  Description: The Turkish validity and reliability of the pain severity scale, originally developed by Price et al. (1994), was established by Eti Aslan (2004) for assessing postoperative pain. This scale, graded from 0 to 10, uses 0 to represent 'I have no pain' and 10 to represent 'I have bearable pain.' Written permission to use the scale was obtained via email from Eti Aslan. A total of Visual Analog Scale (VAS) values were recorded by a study-independent nurse of the study.
State-Trait Anxiety Inventory (STAI) | The first day ; before the blood sugar and insulin procedures and after procedure an average of 1-2 minutes.,
  Description: The State-Trait Anxiety Inventory developed by Spielberger et al. to measure state and trait anxiety levels, was adapted into Turkish by Öner and Le Compte. The STAI-I form was used to assess participants' transitory emotional states and anxiety levels. This 20-item scale utilizes a 4-point Likert scale, with items scored from 1 ('not at all') to 4 ('very much'). The total score, ranging from 20 to 80, indicates anxiety levels, with higher scores signifying greater anxiety. In a Turkish validity and reliability study, the internal consistency coefficients ranged from 0.94 to 0.96. For the current study, the STAI-I's Cronbach's alpha coefficient was determined to be 0.95. The scale was evaluated and recorded by a nurse independent of the study.

SECONDARY OUTCOMES:
Visual analogue scale were used to collect the data. | The second day; during the blood sugar and insulin procedures and , after an average of 1-2 minutes
  The Turkish validity and reliability of the pain severity scale, originally developed by Price et al. (1994), was established by Eti Aslan (2004) for assessing postoperative pain. This scale, graded from 0 to 10, uses 0 to represent 'I have no pain' and 10 to represent 'I have bearable pain.' Written permission to use the scale was obtained via email from Eti Aslan. A total of Visual Analog Scale (VAS) values were recorded by a study-independent nurse of the study.
State-Trait Anxiety Inventory (STAI) | The second day; before the blood sugar and insulin procedures and after an average of 1-2 minutes.
  The State-Trait Anxiety Inventory developed by Spielberger et al. to measure state and trait anxiety levels, was adapted into Turkish by Öner and Le Compte. The STAI-I form was used to assess participants' transitory emotional states and anxiety levels. This 20-item scale utilizes a 4-point Likert scale, with items scored from 1 ('not at all') to 4 ('very much'). The total score, ranging from 20 to 80, indicates anxiety levels, with higher scores signifying greater anxiety. In a Turkish validity and reliability study, the internal consistency coefficients ranged from 0.94 to 0.96. For the current study, the STAI-I's Cronbach's alpha coefficient was determined to be 0.95. The scale was evaluated and recorded by a nurse independent of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Tarsu University, Mersin, Mersin, Health Sciences Faculty ,
  - Tarsus University, Mersin

IPD SHARING:
Plan to Share IPD: No